CLINICAL TRIAL: NCT00158821
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study of the Treatment of Antiretroviral-naive, HIV-1-Infected Patients Comparing Tenofovir Disoproxil Fumarate Administered in Combination With Lamivudine and Efavirenz vs. Stavudine, Lamivudine and Efavirenz.(Extension)
Brief Title: Study of Treatment of Antiretroviral-naive, HIV-1-Infected Patients Comparing Tenofovir Disoproxil Fumarate Administered in Combination With Lamivudine and Efavirenz vs. Stavudine, Lamivudine and Efavirenz.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-99-903; NCT00005573 (obsolete NCT alias)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral; Treatment Experienced; HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; efavirenz; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Viread (tenofovir disoproxil fumarate) — Tenofovir DF 300 mg tablets once daily
  Other Names: Viread
Drug: Sustiva (Efavirenz) — efavirenz capsules 600 mg once daily
  Other Names: Sustiva
Drug: Epivir (Lamivudine) — lamivudine 150 mg tablets twice daily
  Other Names: Epivir
Drug: Zerit (Stavudine) Placebo — stavudine placebo capsules twice daily
  Other Names: Zerit

SUMMARY:
To compare tenofovir DF plus lamivudine plus efavirenz vs. stavudine plus lamivudine plus efavirenz in the treatment of HIV-1-infected patients who have never taken antiretroviral drugs and have a viral load of less than 400 copies/mL at week 48.

DETAILED DESCRIPTION:
To compare the two treatment groups with the goal of achieving HIV-1 RNA levels less than 50 copies/mL at week 48.

To compare the safety, efficacy and tolerability of the two treatment regimens through 144 weeks of drug exposure.

To evaluate the long-term efficacy, safety and tolerability of tenofovir DF in combination with lamivudine and efavirenz through approximately 336 weeks of drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* Completed the original 96-weeks of open-label treatment. Willingness to use effective contraception by both males and females while on study treatment and for 30 days following study drugs completion. The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures related to the second 96-week open-label phase extension.

Exclusion Criteria:

* Patients requiring therapy with any of the following: Nephrotoxic agents (aminoglycoside antibiotics, IV amphotericin B, cidofovir, cisplatin, foscarnet, IV pentamidine, oral and IV vancomycin, oral and IV ganciclovir, other agents with significant nephrotoxic potential);Probenecid; Systemic chemotherapeutic agents; Systemic corticosteroids; Interleukin-2 (IL-2); Investigational agents (except on approval by Gilead Sciences); Drugs that interact with efavirenz (astemizole, terfenadine, dihydroergotamine, ergotamine, midazolam, triazolam, cisapride, rifampin, ergonovine, methylergonovine, voriconazole). Administration of any of the listed medications is not allowed throughout the duration of the study period.
* Pregnant or lactating patients.
* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with patient compliance.
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Patients with biopsy-confirmed cutaneous KS are eligible, if they are not anticipated to require systemic therapy during the study.
* Active, serious infections(other than HIV-1 infection) requiring parenteral antibiotic therapy.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2000-03; Primary Completion 2001-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To compare the two treatment groups with the goal of achieving HIV-1 RNA levels less than 50 copies/mL at week 48. | Week 48
  compare the two treatment groups with the goal of achieving HIV-1 RNA levels
To compare the safety, efficacy and tolerability of the two treatment regimens through 144 weeks of drug exposure. | 144 Weeks
  compare the safety, efficacy and tolerability of the two treatment regimens through 144 weeks of drug exposure

SECONDARY OUTCOMES:
To evaluate the long-term efficacy, safety and tolerability of tenofovir DF in combination with lamivudine and efavirenz through approximately 336 weeks of drug exposure. | 336 Weeks
  evaluate the long-term efficacy, safety and tolerability of tenofovir DF in combination with lamivudine and efavirenz through approximately 336 weeks of drug exposure
To evaluate the long term efficacy, safety and tolerability of tenofovir DF in combination with lamivudine and efavirenz through approximately 480 weeks of drug exposure. | 480 Weeks
  evaluate the long term efficacy, safety and tolerability of tenofovir DF in combination with lamivudine and efavirenz through approximately 480 weeks of drug exposure.
To evaluate the long term efficacy, safety and tolerability of tenofovir DF through approximately 624 weeks of drug exposure. | 624 Weeks
  evaluate the long term efficacy, safety and tolerability of tenofovir DF through approximately 624 weeks of drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: Erin Quirk, M.D., Study Director — Gilead Sciences

REFERENCES:
- [Derived] Madruga JR, Cassetti I, Suleiman JM, Etzel A, Zhong L, Holmes CB, Cheng AK, Enejosa J; Study 903E Team. The safety and efficacy of switching stavudine to tenofovir df in combination with lamivudine and efavirenz in hiv-1-infected patients: three-year follow-up after switching therapy. HIV Clin Trials. 2007 Nov-Dec;8(6):381-90. doi: 10.1310/hct0806-381. PMID 18042503
- See also: Gilead website — http://www.Gilead.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-99-903E_synopsis.pdf